CLINICAL TRIAL: NCT00999986
Title: Phase III Study of the Treatment of Genital Warts by Low Dose Cyclophosphamide
Brief Title: Low Dose Cyclophosphamide Treats Genital Warts
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Feifan Meng, Sheng-Qi-An Biotech Inc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sheng-Qi-An
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Genital Wart
MeSH Terms: conditions — Condylomata Acuminata | interventions — Cyclophosphamide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (No Intervention)
- cyclophosphamide (Active Comparator)
  Interventions: Drug: cyclophosphamide

INTERVENTIONS:
Drug: cyclophosphamide — 50 mg oral per day for 7 days
  Other Names: CY
  Arms: cyclophosphamide

SUMMARY:
Condylomata acuminata (CA) caused by human papillomavirus (HPV) is a common sexually transmitted disease with half a million new cases diagnosed in the United States per year. Recurrence is a major challenge for CA treatment. The investigators have demonstrated that FOXP3+ regulatory T (Treg) cells mediate the immunosuppression in large genital warts. And low-dose cyclophosphamide (CY), a conventional chemotherapy drug, has been reported to selectively deplete Treg cells in cancer patients. Therefore, the investigators hypothesized that low-dose CY can be used to treat genital warts. In this study, 104 CA patients have been recruited for clinical trial with a 1:2 randomization. Among them, 64 patients received low-dose cyclophosphamide and 32 received placebo. In 8 extra patients, high-dose cyclophosphamide was given.

DETAILED DESCRIPTION:
Patients were first treated with CO2 laser therapy, and then treated with low-dose CY, orally 50 mg per day for 7 days.The CA recurrence were observed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of large genital warts

Exclusion Criteria:

* HPV type 6 or 11 was detected negatively by PCR method.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2007-01; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
low-dose cyclophosphamide effectively prevents the recurrence of large genital warts after laser therapy | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Bo Huang, PH.D, MD, Principal Investigator — Tongji Medical College
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

REFERENCES:
- [Background] Cao Y, Zhao J, Lei Z, Shen S, Liu C, Li D, Liu J, Shen GX, Zhang GM, Feng ZH, Huang B. Local accumulation of FOXP3+ regulatory T cells: evidence for an immune evasion mechanism in patients with large condylomata acuminata. J Immunol. 2008 Jun 1;180(11):7681-6. doi: 10.4049/jimmunol.180.11.7681. PMID 18490771
- See also: European Society for Dermatological Research — http://www.esdr.org/index.php?option=com_frontpage&Itemid=1